CLINICAL TRIAL: NCT06688578
Title: Improvements in Balance and Gait Using a Stochastic Noise Stimulator: Short Term Response
Brief Title: Testing Effectiveness of a Stochastic Noise Stimulator to Immediately Improve Balance and Gait
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: University of Western Sydney (Other); National Institute on Aging (NIA) (NIH); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Jorge M. Serrador, Primary Investigator, Massachusetts Eye and Ear Infirmary
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2024P002722; 7R01AG073161 (NIH)
Record Dates: First submitted 2024-11-06; First posted 2024-11-14 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Vestibular Disorder; Aging
Keywords: Balance and Gait; Stochastic Noise Stimulator; Neural degeneration; neuromodulation
MeSH Terms: conditions — Vestibular Diseases; Nerve Degeneration

STUDY DESIGN:
Intervention Model Description: For each test participants will be assessed during stimulation with imperceptible random levels of electrical stimulation as well as during sham stimulation.
Who Masked: Participant, Investigator
Masking Description: Masked individuals will not know if sham or stim;
  1. Participants will be masked.
  2. The Post-doc/Research Coordinator running the study will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham (Sham Comparator): During each testing session there will be a sham and stimulation trial of each test. The order of the sham/stim trials will be randomized.
  Interventions: Device: Sham Comparator
- Stim (Experimental): Three different methods will be used to determine the level of stimulation that produces the greatest improvement in gait. The basic concept is that to determine the optimal level of stimulus the investigators apply various levels of random subperceptual electrical stimulation while measuring either vestibular ocular reflex, static sway or gait. Then the investigators will compare the performance of the selected variable at each level of stimulation to determine which amount of stimulation produced the greatest improvement in the selected variable. Once that is determined
  Interventions: Device: Subperceptual Stimulus

INTERVENTIONS:
Device: Subperceptual Stimulus — For each test participants will be stimulated using a subperceptual electric signal that is optimized to improve their gait.
  Other Names: Novel Treatment of Age-Related Vestibular Loss Using Subperceptual Stimulus
  Arms: Stim
Device: Sham Comparator — During intervention trial, sham comparator will consist of same stimulation device but no actual electrical stimulation will be provided by device during intervention trial.
  Arms: Sham

SUMMARY:
The goal of this intervention study is to determine if a new electronic stimulation device, similar to a TENS can improve balance and make walking easier in older individuals with reduced balance function. The main question aims to answer the following:

Can using the device improve walking speed in older individuals?

Participants will be asked to perform a number of tasks while wearing the device:

Walk for 6 minutes

* Stand in place while having balance measured (eyes open and closed)
* Stand on a foam block while having balance measured (eyes open and closed)
* Sit in a chair that will tilt +/- 20 degrees while wearing goggles that take videos of the participants eyes.

DETAILED DESCRIPTION:
Neural degeneration with age and disease is a recognized and critical problem in health. Despite the significant problems associated with neural degenerative diseases and effects of aging, there remains a lack of effective treatments. An important neural system used daily is the vestibular system. The vestibular system provides continual information on our location in space and is integral to balance, locomotion, daily activities and quality of life. Our lab and others have demonstrated that with increasing age there is a loss of vestibular function that is associated with increased incidence of falls. In fact, falls are the leading cause of injury and death in older Americans (CDC). Older Americans experience 36 million falls per year resulting in 3 million emergency room visits, 700,000 hospitalizations and 32,000 deaths resulting in an estimated $50 billion in annual healthcare costs. Since falls in elderly individuals are associated with greatly increased mortality, reducing fall risk is an essential area to target for healthy aging. Since vestibular function is inherently involved in balance and gait, dealing with age related vestibular loss is an essential component of reducing fall risk. Similarly, patients with vestibular loss have reduced quality of life and increased risk of falls.

Our lab was the first to demonstrate that age related reductions in ocular torsion, a vestibular ocular reflex indicative of otolith function, are associated with increased postural sway in a large group of individuals (N=151) from 21-92 years. Our lab is also the first to demonstrate that subperceptual levels of random electrical stimulation, termed stochastic resonance, are able to improve ocular torsion, indicating improved otolith function, to compensate for age-related vestibular loss.6 Our lab as well as others have also demonstrated that the use of this stimulation can improve static balance and gait in a range of populations. Therefore, a neuromodulation device that could improve balance and gait and reduce fall risk would greatly improve quality of life in aging and reduce mortality. Currently, there are limited treatment options available that can compensate for vestibular loss. A novel neuromodulation treatment is clearly needed. However, current data in this lab and others have only examined the response in the lab over relatively short periods. A recent study found that 3 hours of stimulation improved static balance and this improvement lasted post stimulation for up to 4 hours. These data suggest that this stimulus could be used as a novel rehabilitation device. However there still remains several gaps in knowledge:

1. Do the improvements seen in one system translate to other systems? (i.e., if the investigators see improvement in vestibular ocular reflex, will that translate into improvements in static balance and gait)
2. Do these improvements in static balance translate into gait improvements?

The overall purpose of this study is to investigate whether low level (sub-perceptual) electrical stimulation produces improvements in vestibular function (balance system) that translate into improved balance and gait.

A. Objectives The goal of this study is to determine the cross-modality effectiveness of improving vestibular function on static balance and gait in a population of older individuals with verified reduced vestibular function.

B. Hypotheses / Research Question(s) The overall hypothesis is that stimulation of the vestibular system with extremely low level (subperceptual) electrical signals via surface electrodes will produce immediate improvements in vestibular function that will also translate into improve static balance and gait in older individuals.

ELIGIBILITY:
Inclusion Criteria Older (ages 60+) and younger (aged 21-59) participants with no significant health history will be recruited from the community.

Exclusion Criteria

Any person with a self-reported history of:

* impaired proprioception
* significant eye problems
* neuromuscular disease
* seizure
* stroke
* unmedicated diabetes
* cardiovascular disease (except controlled hypertension)
* renal disease or electrolyte imbalance
* orthopedic disorders such as severe neck or back pain
* uncontrolled high blood pressure (200/110 or greater)
* implanted electronic devices (pacemakers, defibrillators, implanted pumps or stimulator devices, cochlear, etc.)
* psychotic medications or current psychotic symptoms
* Any other psychiatric condition requiring hospitalization since 1991
* recent history of alcohol or drug abuse within the past 6 months
* inability to stand unassisted for 30 seconds or walk unassisted for 6 minutes

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-02-25 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Gait velocity | From enrollment to the end of the intervention (2 days)
  Gait will be measured with a set of motion sensors (Xsens MTw Awinda motion sensors). These wearable inertial monitors measure rotational rate, acceleration, magnetic field strength, and temperature. The sensors are about the size of a watch and attach with Velcro bands. The sensors are wirelessly synchronized with each other and the software, eliminating interconnecting cables and minimizing risk of falling. Gait measures will include gait velocity, gait variability, gait synchronization.

SECONDARY OUTCOMES:
Modified Clinical Test of Sensory Interaction on Balance (mCTSIB) | From enrollment to the end of the intervention (2 days)
  Previous work has demonstrated that posturography provides significant information on vestibular function in the elderly. The mCTSIB will be performed as outlined in the Neurocom geriatric balance assessment to provide an effective initial screening tool. This test involves the subjects standing quietly on a force plate while center of mass and sway are measured with eyes open and closed. To create some instability, subjects will stand quietly on a foam block placed on the force plate with eyes open and then closed. Subjects with poor vestibular function should demonstrate significantly greater sway on tests in which their eyes are closed.
Ocular Torsion | From enrollment to the end of the intervention (2 days)
  OCR is a reflexive torsional eye movement response to a head tilt that has been attributed to the otoliths. It has been demonstrated that OCR is reduced in patients who lack otolithic inputs. Eye movements during OCR tests will be recorded with a videography system that uses the polar cross-correlation technique to measure ocular counter roll using gray scale information of iris patterns obtained from circular sampling paths at fixed radii from the pupil center. To assess otolithic function, binocular counter roll will be recorded with head upright, and then during passive tilting in a chair to the right and left. During the clinical OCR testing portion, the participant will be roll tilted ~30 degrees (whole body) and the eye is measured in roll for both position and velocity.
Video Head Impulse Testing (vHIT) | From enrollment to the end of the intervention (2 days)
  Subject will be fitted with lightweight goggles on which a small camera is mounted. The subject is asked to look at a target while the experimenter gives abrupt horizonal head rotations through a small angle to both the left and the right. The head movement speed is measured by the sensor in the goggles, and the image of the eye is captured by the high-speed camera and processed by very fast software to yield eye velocity. This is a standard clinical vestibular test.
Instrumental Timed Up and Go Test (TUG) | From enrollment to the end of the intervention (2 days)
  Subject will first sit with back against the chair and arms on the armrests. When instructed "Go", the subject will stand up, walk to a marker that is 3 meters away from the chair with their own comfortable and usual speed, and walk back, then sit back down to the chair. Time is taken from the "Go" command until the subject sit back down. This is a standard clinical test for mobility and functional ability with lower times indicate better mobility and lower fall risk.
Functional Gait Assessment (FGA) | From enrollment to the end of the intervention (2 days)
  The FGA is a standard clinical test that usually include 10 walking tasks that assess different aspects of subject's balance and gait. Each task will be scored on a 4-point scale based on the subject's gait quality and stability. A total score from all walking tests will be calculated and higher scores indicate better functional gait performance.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Johns Hopkins Medicine, Baltimore, Maryland
  - Massachusetts Eye and Ear, Harvard Medical School, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
As part of an sIRB agreement, data may be sent to grant research collaborators (Dr. Michael Schubert) at Johns Hopkins School of Medicine to aid in analysis and pursuance of study aims. All data will be de-identified and may include questionnaire results, balance, gait, eye movement data (i.e., OCR and vHIT), and stimulus parameters. Data will be shared with collaborators via current RISO-approved secure methods including REDCap, Veeva, Secure File Transfer, and MGB Dropbox. Clinical data (without any personal identifiers) will be available upon request to the principal investigator (Dr. Jorge Serrador) upon completion of the study.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Upon completion of the study and ending 3 years after the publications of results
Access Criteria: Email the principal investigator (jserrador@meei.harvard.edu)